CLINICAL TRIAL: NCT04571567
Title: A Single-center, Open Label Study to Evaluate the Efficacy and Safety of Secukinumab in Adult Patients With Skin Types IV-VI With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Secukinumab in Adult Patients With Skin Types IV-VI With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saakshi Khattri (Other)
Responsible Party: Sponsor-Investigator, Saakshi Khattri, Assistant Professor, Dermatology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-2408; CAIN457AUS16T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2020-09-26; First posted 2020-10-01 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Skin of Color; Moderate; Severe
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Secukinumab is a recombinant, high-affinity, fully human immunoglobulin G1κ monoclonal antibody targeting IL-17A. Phase III studies have demonstrated the safety and efficacy of secukinumab in the treatment of moderate-to-severe psoriasis when dosed as 300mg by subcutaneous injection at weeks 0, 1, 2, 3, and 4 followed by 300mg every 4 weeks.12 Secukinumab is FDA approved for the treatment of moderate to severe plaque psoriasis in patients 18 years of age and older.
  The study treatment consists of secukinumab 300mg by subcutaneous injection. Each 300mg dose is given as two subcutaneous injections of secukinumab 150mg, 1mg liquid formulation in a pre-filled syringe. Secukinumab pre-filled syringes 150 mg will be supplied by Novartis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Secukinumab (Experimental): 300mg subcutaneously
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Each 300mg dose is given as two subcutaneous injections of secukinumab 150mg, 1mg liquid formulation in a pre-filled syringe.

SUMMARY:
This will be a single-center, open-label clinical study to determine the efficacy and safety of secukinumab in the treatment of moderate to severe psoriasis vulgaris in skin of color (SOC) (FST IV-VI). This study will also evaluate the degree of erythema versus hyperpigmentation in psoriasis plaques in SOC (and its change with secukinumab treatment) as well as the effect of secukinumab on post-inflammatory hyperpigmentation and quality of life in SOC.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disorder primarily affecting the skin and joints that occurs in diverse ethnic groups worldwide. There is paucity of data on the use of topical and systemic medications in dark-skinned individuals. Unique issues in skin of color (SOC) populations, including increased risk of dyspigmentation (hyperpigmentation and hypopigmentation), make studies dedicated to darker skin types essential for treatment of psoriasis in these populations.

This will be a single-center, open-label clinical study to evaluate the efficacy and safety of secukinumab in adults with skin types IV-VI with moderate to severe plaque psoriasis. A total of 20 subjects (ages 18+, male and female, BSA ≥10%, PASI Score ≥ 12, IGA mod 2011 score ≥ 3) are expected to complete this study, which will run for a total of up to 28 weeks.

The study consists of two periods: Screening (from 0 to 4 weeks) and open-label treatment period (24 weeks). During the second period, a total of 20 subjects will receive secukinumab 300mg subcutaneously. Those who meet all of the inclusion/exclusion criteria and are enrolled in the study will receive study drug for the entire treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, signed and dated informed consent prior to initiating any study-related activities.
* Male or female ≥18 years of age at the time of screening
* Fitzpatrick Skin phototype IV-VI, non-white race/ethnicity, including but not limited to African Americans, Asians, Pacific Islanders and Hispanics
* Clinical diagnosis of chronic plaque-type psoriasis of the body for at least 6 months prior to randomization
* Moderate to severe plaque psoriasis at randomization as defined by: PASI≥12 AND BSA ≥ 10% AND IGA mod 2011 ≥ 3 (scale 0-4)
* Candidate for systemic therapy, as defined by having psoriasis inadequately controlled by topical treatments and/or phototherapy and/or previous systemic therapy
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While using investigational product and for at least 28 days after last application of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below: Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
* Must be in general good health as judged by the Investigator, based on medical history and physical examination. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).

Exclusion Criteria:

* Form of diagnosed psoriasis other than chronic plaque psoriasis (i.e. guttate, erythrodermic, pustular) or drug-induced psoriasis
* Subjects with lighter skin as defined by Fitzpatrick Skin Types I-III
* Subjects of European ancestry or other white ethnic group
* Previous exposure to secukinumab or other biologic agent targeting IL-17A or IL-17RA
* Ongoing use of prohibited treatments or lack of adherence to specified washout periods:

  * 6 months for biologic drugs directly targeting IL-12/23 or IL-23, alefacept, and efalizumab
  * 12 weeks for biologic agents other than the above (i.e. adalimumab, etanercept, infliximab)
  * 4 weeks for other systemic psoriasis treatments (i.e. methotrexate, systemic steroids, retinoids, apremilast), and photochemotherapy
  * 2 weeks for phototherapy (UVA, UVB)
  * 2 weeks for topical psoriasis therapies
* Subjects unwilling to limit exposure to UV light
* Use of other investigational drugs within 5 half-lives prior to randomization
* Pregnant/nursing women or women of child-bearing potential unwilling to use appropriate method of contraception
* Diagnosis of other ongoing skin disease or skin infection that may interfere with the treatment and/or examination of psoriasis lesions
* Current significant medical problems or laboratory abnormalities that, in the opinion of the investigator, would put the patient at significant risk by participating in the study
* Previous history of or current infection with hepatitis C, hepatitis B, or HIV
* Active systemic infection during the 2 weeks prior to randomization
* Evidence of tuberculosis infection (indeterminate or positive quantiferon gold) at screening. Subject may be enrolled if full tuberculosis workup has been completed in the 12 weeks preceding randomization and patient has been started on appropriate treatment at least 4 weeks prior to randomization
* Malignancy with the past 5 years, with the exception of basal cell carcinoma, actinic keratosis, Bowen's disease of the skin, carcinoma in situ of the cervix(removed) or non-invasive malignant color polyps (removed)
* History of allergy to any component of the IP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Psoriasis Area Severity Index (PASI) 90 | Baseline, Week 16 and Week 24
  Proportion of patients achieving ≥90% improvement in Psoriasis Area Severity Index (PASI) at week 16 compared to baseline (PASI90). PASI will be assessed at baseline and then at regular intervals until week 24.

SECONDARY OUTCOMES:
Change in PASI 75 | Baseline, Weeks 4, 12, 16, and 24
  PASI 75 at weeks 4, 12, 16, 24 - Proportion of patients achieving ≥75% improvement in Psoriasis Area Severity Index (PASI) at weeks 4, 12, 16, and 24 compared to baseline (PASI75).
Change in PASI 90 | Baseline, Weeks 4, 12, 16, and 24
  PASI 90 at weeks 4, 12, 24 - Proportion of patients achieving ≥90% improvement in Psoriasis Area Severity Index (PASI) at weeks 4, 12, and 24 compared to baseline (PASI90).
Change in PASI 100 | Baseline, Weeks 4, 12, 16, and 24
  PASI 100 at weeks 4, 12, 16, 24 - Proportion of patients achieving 100% improvement in Psoriasis Area Severity Index (PASI) at weeks 4, 12, 16, and 24 compared to baseline (PASI100).
Change in Investigator Global Assessment (IGA) mod 2011 | Weeks 12, 16, and 24
  IGA mod 2011 0/1 at weeks 12, 16, 24 - Proportion of patients at weeks 12, 16, and 24 who achieved treatment success according to investigator global assessment (IGA mod 2011) of the entire body including scalp. IGA full range from 0 (clear) to 4 (severe). Treatment success is defined as IGA of clear (0) or almost clear (1).
Change in The Physician Global Assessment and Body Surface Area (PGAxBSA) score | Baseline and Week 16
  ≥75% reduction in IGAxBSA score (IGAxBSA-75) at week 16 - ≥75% improvement in PGAxBSA Composite Tool between week 16 and baseline. The PGAxBSA score is calculated by multiplying the static PGA score by the BSA (range: 0 to 400 [eg, maximum static PGA = 4 and maximum BSA = 100]).
Change in melanin index (MI) | Weeks 4, 12, 16, 24
  Change in melanin index (MI) of target lesion at weeks 12, 16, 24 compared to week 4. Melanin index total scale from 0-999, higher score indicates higher melanin content.
Change in erythema index (EI) | Baseline, Weeks 4, 12, 16, and 24
  A skin spectrophotometer (Mexameter) will be used to quantify the MI (degree of hyperpigmentation or hypopigmentation) and EI of lesional skin compared to an index area of unaffected skin at baseline, week 4, week 12, week 16, and week 24 as compared to baseline. Full scale from 0-4, higher score indicates more erythema
Change in physician numeric rating scale (physician) | Baseline, Weeks 4, 12, 16, and 24
  The physician dyspigmentation NRS ranges from 5 (severe dark brown pigmentation) to -5 (complete absence of pigment), with 0 being baseline skin pigmentation. The scale is as follows: 5 severe dark brown pigmentation (darkest imaginable color), 4 dark brown pigmentation, 3 medium brown pigmentation, 2 light brown pigmentation, 1 slight dark pigmentation (barely perceptible compared to surrounding skin), 0 baseline skin pigmentation, -1 slight hypopigmentation (barely perceptible compared to surrounding skin), -2 mild hypopigmentation (light brown), -3 moderate hypopigmentation (creme-colored skin), -4 severe hypopigmentation (almost complete absence of pigment), -5 depigmentation (complete absence of pigment). Only one number along the scale will be chosen (corresponding to either hypopigmentation or hyperpigmentation). Change at weeks 12, 16, and 24 compared to Week 4.
Change in patient-rated visual analog scale | Baseline, Weeks 4, 12, 16, and 24
  The NRS ranges from 5 (severe dark brown pigmentation) to -5 (complete absence of pigment), with 0 being baseline skin pigmentation. The scale is as follows: 5 severe dark brown pigmentation (darkest imaginable color), 4 dark brown pigmentation, 3 medium brown pigmentation, 2 light brown pigmentation, 1 slight dark pigmentation (barely perceptible compared to surrounding skin), 0 baseline skin pigmentation, -1 slight hypopigmentation (barely perceptible compared to surrounding skin), -2 mild hypopigmentation (light brown), -3 moderate hypopigmentation (creme-colored skin), -4 severe hypopigmentation (almost complete absence of pigment), -5 depigmentation (complete absence of pigment). Only one number along the scale will be chosen (corresponding to either hypopigmentation or hyperpigmentation). Change at weeks 12, 16, and 24 compared to Week 4.
Change in the Dermatology Life Quality Index (DLQI) | Weeks 12, 16, and 24
  Change from baseline in DLQI total score and proportion of subjects achieving DLQI 0/1 at weeks 12, 16, 24. Full scale from 0-10, with higher score indicating more impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Saakshi Khattri, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West Dermatolgy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data.To achieve aims in the approved proposal.OtherUnknown at this time.